CLINICAL TRIAL: NCT06976190
Title: A Randomized, Open-label, Multi-center, Phase III Study of MRG003 in Combination With Pucotenlimab Versus Chemotherapy in the Treatment of Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma
Brief Title: A Study of MRG003 in Combination With Pucotenlimab Versus Chemotherapy in the Treatment of Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma
Acronym: Magic-C002
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HX008/MRG003-C002
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Recurrent or Metastatic Nasopharyngeal Carcinoma
Keywords: MRG003; Pucotenlimab; Nasopharyngeal Carcinoma
MeSH Terms: conditions — Recurrence; Nasopharyngeal Carcinoma | interventions — Gemcitabine; Docetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRG003 + Pucotenlimab (Experimental)
  Interventions: Drug: MRG003 + Pucotenlimab
- Chemotherapy Arm (Active Comparator): Mono-chemotherapy as selected by investigator
  Interventions: Drug: Gemcitabine, Docetaxel, or Capecitabine

INTERVENTIONS:
Drug: MRG003 + Pucotenlimab — MRG003 will be administrated as specified in the protocol. Pucotenlimab will be administrated as specified in the protocol.
  Arms: MRG003 + Pucotenlimab
Drug: Gemcitabine, Docetaxel, or Capecitabine — Gemcitabine will be administrated via intravenous infusion at 1000 mg/m2 once on Day 1 and 8 of every 3 weeks (21-day cycle).
  Docetaxel will be administrated via intravenous infusion at 75 mg/m2 once on Day 1 of every 3 weeks (21-day cycle).
  Capecitabine will be administrated orally at 1000 mg/m2 twice a day for Day 1 to 14 of every 3 weeks (21-day cycle).
  Arms: Chemotherapy Arm

SUMMARY:
This is a randomized, open-label, multi-center, phase III study to evaluate the efficacy and safety, and immunogenicity of MRG003 in combination with pucotenlimab in patients with recurrent or metastatic nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign the informed consent form and follow the requirements specified in the protocol.
* Life expectancy ≥ 12 weeks.
* Patients with histologically and cytologically confirmed recurrent or metastatic nasopharyngeal carcinoma (NPC) who have failed at least one line of prior systemic therapy.
* Patients must have at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
* The score of ECOG for performance status is 0 or 1.
* No severe cardiac dysfunction, left ventricular ejection fraction (LVEF) ≥50%.
* Organ functions and coagulation function must meet the basic requirements.
* Patients with childbearing potential must use effective contraception during the treatment and for 6 months after the last dose of treatment.

Exclusion Criteria:

* History of hypersensitivity to any component of the investigational product.
* Received systemic chemotherapy, targeted therapy, biological therapy or immunotherapy for anti-tumor purpose, or major surgery within 3 weeks prior to the first dose of study treatment.
* Received anti-infection therapy within 2 weeks prior to the randomization
* Prior treatment with MMAE/MMAF ADC drugs
* Central nervous system metastasis.
* Poorly controlled systemic diseases
* Patients with poorly controlled heart diseases
* Poorly controlled pleural and peritoneal effusion or pericardial effusion
* ≥Grade 2 toxic reaction or abnormal value of laboratory test caused by previous anti-tumor treatment
* Patients with prior ≥Grade 3 immuno-related adverse events (irAEs)
* Any clinically significant arteriovenous bleeding, pulmonary embolism, or deep venous thrombosis occurred within 3 months
* Received allogeneic tissue/solid organ transplantation.
* Inoculate live vaccine within 30 days before the first dose.
* Patients with a positive serum pregnancy test or who are breast-feeding or who do not agree to take adequate contraceptive measures during the treatment and for 180 days after the last dose of study treatment.
* History of other primary malignant tumor diseases.
* Other situations that are not suitable to participate a clinical trial per investigator's judgement

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) as assessed by BIRC | Baseline to study completion (up to 33 months)
  PFS is defined as the duration from the start of treatment to the onset of tumor progression or death of any cause.
Overall Survival (OS) | Baseline to study completion (up to 48 months)
  OS is defined as the duration from the start of treatment to death of any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Baseline to study completion (up to 48 months)
  ORR is defined as the proportions of patients with a complete response (CR) and partial response (PR). ORR will be assessed according to RECIST v1.1.
Disease Control Rate (DCR) | Baseline to study completion (up to 48 months)
  DCR is defined as the proportion of subjects achieving CR, PR, and stable disease (SD) after treatment.
Progression Free Survival (PFS) as assessed by investigator | Baseline to study completion (up to 33 months)
  PFS is defined as the duration from the start of treatment to the onset of tumor progression or death of any cause.
Immunogenicity (ADA) | Baseline to 14 days after the last dose.
  The proportion of patients with positive ADA results.
Adverse Events (AEs) | Baseline to 30 days after the last dose of study treatment
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial whether or not the event is considered related to the study drug.
Serious Adverse Events (SAEs) | Baseline to 30 days after the last dose of study treatment
  Adverse events that are fatal, life-threatening, or result in hospitalization or prolonged hospitalization, persistent or significant disability/incapacity/substantial disruption of the ability to lead a normal life, congenital anomaly/birth defect or major medical events or reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No